CLINICAL TRIAL: NCT03980236
Title: Feasibility of Using the Insulia App in an Integrated Platform With Livongo for Patients With Type 2 Diabetes Treated With Basal Insulin [Pilot Study]
Brief Title: Feasibility of Using the Livongo-Insulia Study App for Patients With Type 2 Diabetes [Pilot Study]
Acronym: LISA Pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not achieve enrollment goal
Sponsor: Livongo Health (Industry)
Collaborators: Voluntis (Industry); Evidation Health (Industry)
Responsible Party: Principal Investigator, Bimal Shah, MD, Co-Principal Investigator, Livongo Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CP04573.A
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes Treated With Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Livongo-Insulia Study App Arm (Experimental): Participants will be asked to use the Livong-Insulia Study App for the 3 month study duration
  Interventions: Device: Livongo-Insulia Study App

INTERVENTIONS:
Device: Livongo-Insulia Study App — Throughout the study, participants will be asked to use the LIvongo-Insulia Study App daily to receive their basal insulin dose recommendation. Participants will need to check their before breakfast blood glucose using their Livongo meter. Then, they will need to open the Livongo-Insulia Study App and accept the uploaded blood glucose(s) from the Livongo meter. Once the appropriate information is received, participants will receive an insulin dose recommendation and should confirm once the dose has been taken. Depending on their blood glucose, participants may also receive coaching messages and coaching support from the Livongo program.

SUMMARY:
The Livongo-Insulia Study App Pilot Study (LISA Pilot) is a 3-month, prospective, interventional study. The purpose of this pilot study is to evaluate the feasibility of using the Livongo-Insulia Study App for individuals with type 2 diabetes using basal insulin. This will be assessed by measuring the impact of the Livongo-Insulia Study App on glycemic control for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Lives in the U.S.
* Able to speak, read and write in English
* Diagnosed with type 2 diabetes
* Currently treated with long-acting basal insulin analog (Lantus, Levemir, Toujeo, Basaglar, Tresiba U-100) and taking 1 injection per day
* Takes a daily dose ≤ 0.75 units/kg
* Estimated A1c ≥ 8% (based on existing Livongo data)
* Has been enrolled in Livongo for at least 12 weeks
* Uses an iPhone compatible with Insulia's compatibility matrix (iPhone 5 or higher; iOS 8 or newer)
* Willing to complete study questionnaires
* Willing to complete at-home A1c kits
* Willing to check before breakfast blood glucose at least once per day

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Currently using a long-acting basal insulin analog that is not supported by Insulia
* Currently using rapid-acting, short-acting, or intermediate-acting or premixed insulins
* Currently pregnant or planning pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in A1c | 12 weeks
  Change in A1c from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bimal Shah, MD, MBA, Principal Investigator — Livongo Health
Locations (1):
- Livongo, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No